CLINICAL TRIAL: NCT03037619
Title: Influence of Wearable Activity Monitors and Social Support on Physical Activity After Knee Replacement
Brief Title: Fitbit and Social Support in Knee Replacement Patients & Buddies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Christine A Pellegrini, PhD, Research Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00063842
Record Dates: First submitted 2017-01-27; First posted 2017-01-31 (Estimated); Results first posted 2019-09-16 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fitbit (Experimental): Participants randomized to Fitbit will be mailed a Fitbit and encouraged to wear it over the next 4 months.
  Interventions: Behavioral: Fitbit
- Fitbit+Support (Experimental): Participants will identify a Buddy and both the participant and Buddy will be mailed a Fitbit. Both participant and Buddy will be asked to "Friend" each other on Fitbit and encouraged to wear the monitor over the next 4 months.
  Interventions: Behavioral: Fitbit+Support

INTERVENTIONS:
Behavioral: Fitbit — Participants randomized to Fitbit will be mailed a Fitbit and encouraged to wear it over the next 4 months
  Arms: Fitbit
Behavioral: Fitbit+Support — Participants will identify a Buddy and both the participant and Buddy will be mailed a Fitbit. Both participant and Buddy will be asked to "Friend" each other on Fitbit and encouraged to wear the monitor over the next 4 months.
  Arms: Fitbit+Support

SUMMARY:
Patients undergoing knee replacement typically report improved health-related quality of life, increased physical function, and reduced pain. Despite these improvements, physical activity levels remain unchanged, or only minimally increase from pre-operative levels, yet do not reach the same level of activity observed among healthy populations. Knee replacement patients often expect their activity levels and function to improve following surgery, but the majority of patients' activity levels 5 years post-operatively did not meet their pre-operative expectations. Even though improvements are observed in pain and function, reasons for the maintenance of low levels of activity are unknown. Technology has the potential to increase physical activity levels in these patients, particularly as 81% of knee replacement patients in our recent study had a smartphone, and 40% were willing to wear a wrist-worn physical activity monitor. As the average age of knee replacement continues to decrease, we anticipate that the percent of patients with a smartphone and willingness to wear an activity monitor will increase. In addition to technology, social support is associated with greater outcomes following knee replacement. Thus, wearing a wrist-worn physical activity monitor and providing additional opportunities for social support via the technology may increase physical activity levels in these patients. The current pilot study aims to gain preliminary data on the influence of wearables and social support on physical activity in knee replacement patients following surgery. Specifically, we aim to recruit 20 patients who will be randomized to one of two conditions: Fitbit vs. Fitbit+Support. Participants in the Fitbit group will receive a Fitbit and be encouraged to wear it for 4 months. Participants in the Fitbit+Support group will be asked to identify a "buddy." Both the participant and "buddy" will be given a Fitbit and they will be asked to friend each other via Fitbit and wear the monitor for 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Knee replacement patients must (1) have had a knee replacement in the last 12 months; (2) have a computer or smartphone compatible with Fitbit, (3) be English speaking, (4) willing to wear the Fitbit for 4 months, and (5) have a "buddy" willing to participate.
* Patient buddies must: (1) have a computer or smartphone compatible with Fitbit, (2) be English speaking, and (3) willing to wear the Fitbit for 4 months.

Exclusion Criteria:

* Knee replacement patients will be excluded if they have another knee replacement scheduled within the next 4 months.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2018-11-10 (Actual); Study Completion 2018-11-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fitbit | Fitbit+Support
Started | 8 | 15 (8 participants and 7 buddies)
Completed | 8 | 14 (7 participants and 7 buddies)
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: "Buddy participants" (n=7) were excluded from baseline analyses. Only knee replacement participants were included (n=8).
Groups:
- Fitbit&Support: Participants will identify a Buddy and both the participant and Buddy will be mailed a Fitbit. Both participant and Buddy will be asked to "Friend" each other on Fitbit and encouraged to wear the monitor over the next 4 months.
  Fitbit+Support: Participants will identify a Buddy and both the participant and Buddy will be mailed a Fitbit. Both participant and Buddy will be asked to "Friend" each other on Fitbit and encouraged to wear the monitor over the next 4 months.
- Total: Total of all reporting groups
Arm/Group | Fitbit | Fitbit&Support | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 4 | 10
  >=65 years | 2 | 4 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (7.6) | 62.5 (8.5) | 60.6 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 0 | 3 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8

OUTCOME MEASURES:

1. Primary Outcome: Moderate/Vigorous Intensity Physical Activity
Description: Number of minutes/day of moderate and vigorous intensity physical activity measured by the Fitbit
Time Frame: 4 months
Population: "Buddy participants" (n=7) were excluded from Fitbit+Support main analyses. Only knee replacement participants who completed the study were included in analyses
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Fitbit | Fitbit+Support
Number analyzed (Participants) | 8 | 7
minutes/day | 26.9 (28.4) | 33.1 (32.7)

2. Secondary Outcome: Social Support
Description: Social Support & Exercise Survey - Family score (sum items 11 - 16 and 20 - 23); Scores can range between 10-50, with a higher score indicating more support
Time Frame: 4 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fitbit | Fitbit+Support
Number analyzed (Participants) | 8 | 7
score on a scale | 16.6 (7.9) | 25.0 (12.2)

3. Secondary Outcome: Percentage of Participants Satisfied With the Fitbit
Description: Acceptability of the Fitbit (% satisfied with Fitbit)
Time Frame: 4 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fitbit | Fitbit+Support
Number analyzed (Participants) | 8 | 7
Participants | 7 | 6

4. Secondary Outcome: Fitbit Engagement
Description: Percentage of days Fitbit was worn
Time Frame: 4 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Fitbit | Fitbit+Support
Number analyzed (Participants) | 8 | 7
Percentage of days | 88.9 (13.2) | 99.3 (1.3)

ADVERSE EVENTS:
Time Frame: 4 months
Description: This study was classified as minimal risk to participants.
Arm/Group | Fitbit | Fitbit+Support
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/15
Other Adverse Events (participants affected / at risk) | 0/8 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-21): https://cdn.clinicaltrials.gov/large-docs/19/NCT03037619/Prot_SAP_000.pdf